CLINICAL TRIAL: NCT03115879
Title: The Effect of High Velocity Low Amplitude Hip Mobilization on Strength in Subjects With Lower Extremity Pathology
Brief Title: The Effect High Velocity Low Amplitude Hip Mobilization on Strength in Subjects With Lower Extremity Pathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Diego Galace de Freitas, Principal Investigator, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DFreitas
Record Dates: First submitted 2017-03-23; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Hip Joint; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Hip manipulation simulation
  Interventions: Other: Hip manipulation simulation
- Manipulation Group (Experimental): Hip manipulation
  Interventions: Other: Hip mobilization

INTERVENTIONS:
Other: Hip mobilization — High velocity low amplitude hip mobilization of the experimental group
  Arms: Manipulation Group
Other: Hip manipulation simulation — Hip manipulation simulation
  Arms: Placebo Group

SUMMARY:
Introduction: Lower extremity weakness associated with musculoskeletal pathology can cause activity limitations. Physical therapy intervention in the form of exercise is commonly directed at improving muscular performance, however, neuromuscular adaptations may limit the effectiveness of traditional strengthening exercises. Manual therapy techniques have been used as a disinhibitory intervention to increase muscle activation and strength before participating in strengthening exercises or performing functional tasks While there is recent evidence to support joint mobilization as a valuable manual therapy disinhibitory intervention Currently, there is no evidence to substantiate anecdotal experience that a HVLAT hip distraction mobilization improves muscle performance in subjects with lower extremity pathology and lower extremity weakness. The purpose of this study was to determine if a HVLAT hip distraction mobilization would result in an immediate change of maximal force output of the quadriceps, gluteus maximus and gluteus medius.

Methods: Forty individuals with a lower extremity pathology volunteered for this study. Inclusion criteria were having a unilateral musculoskeletal pathology, being greater than 18 years of age, 10% decrease in muscle strength in symptomatic side compared to healthy side, and absence of medical precautions that would prevent a maximal effort strength test and exclusion criteria included individuals with a history lower extremity recent muscle or tendon ruptures (within the past 6 months) and postoperative knee, hip and ankle surgery. Demographic data, including diagnosis from referring physician were collected. All subjects completed the Lower extremity function scale (LEFS). A single evaluator blinded to the involved extremity was responsible for quadriceps, gluteus medius and maximus strength analysis pre and post mobilization of both symptomatic and non-symptomatic sides. The subject underwent the HVLAT hip distraction mobilization of the symptomatic side, and an immediate re-assessment of strength of both symptomatic and non-symptomatic sides followed the mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a lower extremity pathology volunteered for this study
* Being greater than 18 years of age
* 10% decrease in muscle strength in symptomatic side compared to healthy side
* Absence of medical precautions that would prevent a maximal effort strength test.

Exclusion Criteria:

* Included individuals with a history lower extremity arthroplasty.
* Recent muscle or tendon ruptures (within the past 6 months)
* Unhealed fractures
* Neurological diseases
* Malignant cancer
* Osteoporosis
* Active infections processes
* Early postoperative knee, hip and ankle surgery with range of motion and weight bearing restrictions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Muscle strength | Assessment of muscle strength was performed after 10 minutes of manipulation
  A Lafayette dynamometer was used to evaluate the maximum isometric torque of the muscles